CLINICAL TRIAL: NCT03438721
Title: Strong Futures: A Pilot Randomized Controlled Trial of Two Primary Care Based Interventions to Promote Optimal Health in Latino Infants and Toddlers
Brief Title: Strong Futures: A Trial of Two Primary Care Based Interventions to Promote Optimal Health in Latino Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-24028; 1K23HD080876-01A1 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-02-20 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Childhood Obesity; Health-Related Quality of Life
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant Obesity Prevention (Experimental): The infant obesity prevention arm will provide parents with education on optimal infant feeding, sleep, and screen time practices.
  Interventions: Behavioral: Infant obesity prevention
- Financial Coaching (Experimental): The financial coaching arm will provide parents with education on basic financial literacy topics and coaching to help parents achieve financial goals.
  Interventions: Behavioral: Financial coaching

INTERVENTIONS:
Behavioral: Infant obesity prevention — Parents will receive education on infant feeding, sleep, and screen time practices just after well-child visits in the first year of life. The education will be provided by a lay health educator. Parents will also receive text messages to reinforce the intervention content
  Arms: Infant Obesity Prevention
Behavioral: Financial coaching — Parents randomized to the financial coaching arm will receive basic education on financial topics including budgeting, savings, and managing debt as well as coaching on these topics just after well-child visits in the first year of life. Coaching will be provided by lay health educators trained in financial coaching. Parents will also receive text messages reinforcing the information learned.
  Arms: Financial Coaching

SUMMARY:
Latino children experience higher rates of obesity compared to non-Hispanic white children, especially in low-income communities. Optimal feeding strategies in early life, avoidance of screen time and longer sleep duration may lower the risk of obesity. Family financial hardship is also associated with short- and long-term health risks, including behavioral and mental health problems, and toxic stress which contributes to elevated risk of common chronic conditions over the life course. This proposal aims to pilot test two interventions to promote optimal health outcomes in Latino infants. Study participants will meet with a health educator after well child visits at 2-weeks, 2-, 4-, 6-, 9- and 12-months. Half of the parents will receive education on obesity prevention. The other half will receive financial education and case management using an established financial coaching approach. Parents will also receive text messages that reinforce educational content. The objective of this study is to determine the acceptability and feasibility of offering these interventions in the well-child setting. Study investigators also seek to determine the preliminary efficacy of these interventions on infant and parent health outcomes including dietary intake, screen time, sleep duration, health related quality of life and financial stress.

ELIGIBILITY:
Inclusion Criteria:

* Study investigators will recruit parents who self-identify as Latino and their newborn infants
* Infants must be born at Zuckerberg San Francisco General Hospital (ZSFG)
* Infants must be singletons
* Parents must intend to receive primary care for their infant at Zuckerberg San Francisco General Hospital
* Parents must speak Spanish (but may also speak English)

Exclusion Criteria:

* Infants with birth weights less than 2500 grams
* Infants born prior to 37 weeks and 0 days gestation
* Infants with any medical condition that significantly affects feeding, such as infants who are unable to feed by mouth
* Infants with any medical condition that is known to be associated with failure to thrive or specialized nutritional needs
* Infants in foster care
* Infants for whom the primary caregiver is not the infant's mother or father

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Child dietary intake | 15-months
  Total child intake of sugar-sweetened-beverages and 100% fruit juice in ounces and total intake of fruits and vegetables in grams.
Child screen time | Child age 15-months
  Total minutes of daily screen time
Parent health-related quality of life | Child age 15-months
  Assessed by the PROMIS-10. The Patient Reported Outcome Measurement Information System Global Short Form 10 (PROMIS-10) is a ten-item scale measuring health related quality of life with subscales for physical and mental health. Raw overall total PROMIS-10 scale scores range from 10-50, with sub-scale T-scores that range from 16-67 for physical health and 21-68 for mental health. For all PROMIS-10 total raw and sub-scale scores, higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Child anthropometrics | Child ages 6-months, 12-months, 15-months and 24-months
  World Health Organization Weight-for-length z-score
Parent financial stress | Child age 15-months
  Consumer Financial Protection Bureau Financial Well-Being Scale. The Consumer Financial Protection Bureau Financial Well Being Questionnaire (Short Form, CFPB Financial Well Being Questionnaire SF) is a five item scale measuring individual financial well-being. The CFPB Financial Well Being Questionnaire has a range of 0-20 raw score, based on a 5-point Likert scale for each item, with one item (item 4) reverse coded and summed with responses for the remaining items to arrive at the raw score. The raw score is converted to a reference financial well-being score.Higher scores indicate greater financial well-being.
Child sleep | Child age 15-months
  Child total minutes of sleep in 24-hour period
Parental feeding styles | 15-months
  Study investigators will assess responsive, pressuring and indulgent feeding styles using the "responsive satiety," "pressuring finishing," "pressuring soothing," and "indulgence permissive" sub-scales of the Infant Feeding Styles Questionnaire. These sub-scales assess both behaviors and beliefs relevant to the construct. Scores range from 1-5 with higher scores indicating greater use of that feeding style.

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Beck, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Children's Health Center at San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No